CLINICAL TRIAL: NCT00702156
Title: Cardioselective Beta-Blockade Using Bisoprolol in Patients With Chronic Heart Failure (CHF) and Coexistent Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD) With or Without Significant Reversibility.
Brief Title: Bisoprolol in Patients With Heart Failure and Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patient recruitment
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Dr Nathaniel Hawkins, Glasgow Royal Infirmary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RN05CA013
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-08

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Heart Failure; Chronic Obstructive Pulmonary Disease; Beta-blockers; Pulmonary Function
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bisoprolol
  Interventions: Drug: Bisoprolol
- 2 (Placebo Comparator): Identical appearance matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol — Titration. 1.25 mg 2 weeks, 2.5 mg 2 weeks, 5 mg 4 weeks, 7.5 mg 4 weeks, 10 mg 4 weeks.
  Other Names: Bisoprolol Fumarate; Brand name: Cardicor
  Arms: 1
Drug: Placebo — Titration. 1.25 mg 2 weeks, 2.5 mg 2 weeks, 5 mg 4 weeks, 7.5 mg 4 weeks, 10 mg 4 weeks.
  Arms: 2

SUMMARY:
The principal research objectives are to demonstrate cardioselective beta-blockade using bisoprolol is not inferior to placebo with regard to pulmonary function and improves quality of life in patients with heart failure and coexistent moderate or severe chronic obstructive pulmonary disease with or without significant reversibility. Patients will be followed up for 4 months during which bisoprolol will be up-titrated to the maximum clinically tolerated dose. Health status will be assessed using a generic and two disease specific questionnaires, and pulmonary function by spirometry, body box plethysmography, and cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic NYHA II or III chronic heart failure
* left ventricular systolic dysfunction
* moderate or severe chronic obstructive pulmonary disease
* with or without significant reversibility

Exclusion Criteria:

* beta-blocker contraindications
* non-dihydropyridine (diltiazem / verapamil) calcium channel blockers
* recent coronary percutaneous intervention or coronary artery bypass graft surgery
* haemodynamically significant valvular disease or hypertrophic cardiomyopathy.
* active myocarditis or pericarditis.
* recent cerebrovascular accident or transient ischaemic attack
* serious concurrent systemic disease, such as malignancy, resulting in likely reduced life expectancy
* pregnancy, childbearing potential with inadequate contraception, breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-03; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume 1 second (FEV1) | 16 weeks

SECONDARY OUTCOMES:
Quality of life: Minnesota Living with Heart Failure, SF-36 | 16 weeks
NYHA Class | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel M Hawkins, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde; Francis G Dunn, MBChB MD, Study Chair — NHS Greater Glasgow and Clyde; Roger Carter, BSc MSc PHD, Study Director — NHS Greater Glasgow and Clyde; George W Chalmers, MBChB MD, Study Director — NHS Greater Glasgow and Clyde
Locations (1):
- Cardiopulmonary Transplant Unit Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Hawkins NM, MacDonald MR, Petrie MC, Chalmers GW, Carter R, Dunn FG, McMurray JJ. Bisoprolol in patients with heart failure and moderate to severe chronic obstructive pulmonary disease: a randomized controlled trial. Eur J Heart Fail. 2009 Jul;11(7):684-90. doi: 10.1093/eurjhf/hfp066. Epub 2009 May 21. PMID 19460848